CLINICAL TRIAL: NCT03601806
Title: A Phase II Multicenter Study of Pomalidomide Monotherapy in HIV-Positive Individuals With Kaposi Sarcoma (KS) in Sub-Saharan Africa (SSA)
Brief Title: Pomalidomide in Treating Patients With Kaposi Sarcoma and Human Immunodeficiency Virus Infection
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: AIDS Malignancy Consortium (Network)
Collaborators: National Cancer Institute (NCI) (NIH); The Emmes Company, LLC (Industry); University of Arkansas (Other); Montefiore Medical Center (Other); University of Stellenbosch (Other); Weill Medical College of Cornell University (Other); University of California, Los Angeles (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AMC-100; NCI-2017-00390 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); AMC-100; AMC-100 (Other: AIDS Malignancy Consortium); AMC-100 (Other: CTEP); UM1CA121947 (NIH)
Record Dates: First submitted 2018-07-18; First posted 2018-07-26 (Actual); Results first posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-12

CONDITIONS: Human Immunodeficiency Virus 1 Positive; Skin Kaposi Sarcoma
MeSH Terms: interventions — pomalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Treatment (pomalidomide) (Experimental): Patients receive pomalidomide PO QD on days 1-21. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.
  Interventions: Other: Laboratory Biomarker Analysis; Drug: Pomalidomide

INTERVENTIONS:
Other: Laboratory Biomarker Analysis — Correlative studies
Drug: Pomalidomide — Given PO
  Other Names: 4-Amino thalidomide; Actimid; CC-4047; Imnovid; Pomalyst

SUMMARY:
This phase II clinical trial studies the side effects of pomalidomide and how well it works in treating patients with Kaposi sarcoma and human immunodeficiency virus (HIV) infection. Biological therapies, such as pomalidomide, may stimulate the immune system in different ways and stop tumor cells from growing and it may also block the growth of new blood vessels necessary for tumor growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine if pomalidomide monotherapy induces a minimal level of antitumor efficacy to justify its further development for HIV-associated Kaposi sarcoma (KS) in sub-Saharan Africa and is safe and tolerable.

SECONDARY OBJECTIVES:

I. To evaluate the effects of pomalidomide monotherapy on standard measures of HIV control, i.e., CD4 counts and HIV viral loads, in this participant population.

TERTIARY OBJECTIVES:

I. To assess the effect of pomalidomide treatment on serum cytokine levels. II. To evaluate if changes in serum cytokine levels correlate with clinical response.

OUTLINE:

Patients receive pomalidomide orally (PO) once daily (QD) on days 1-21. Treatment repeats every 28 days for up to 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 12 weeks for 48 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Participants must have measurable cutaneous KS that has been pathologically confirmed by an acquired immunodeficiency syndrome (AIDS) Malignancy Consortium (AMC)-approved pathologist; diagnostic tissue must be available to satisfy the tissue submission requirements for central pathology review
* Participants may not show evidence for ongoing improvement in KS lesions in the 4 weeks prior to enrollment
* HIV positive. Documentation of HIV-1 infection by means of any one of the following:
* HIV-1 RNA detection by a licensed HIV-1 RNA assay demonstrating >1000 RNA copies/mL confirmed by a licensed screening antibody and/or HIV antibody antigen combination assay;
* Any licensed HIV screening antibody and/or HIV antibody/antigen combination assay confirmed by a second licensed HIV assay such as a HIV-1 Western blot confirmation or HIV rapid multispot antibody differentiation assay. NOTE: The term "licensed" refers to a kit that has been certified or licensed by an oversight body within the participating country and validated internally. WHO (World Health Organization) and CDC (Centers for Disease Control and Prevention) guidelines mandate that confirmation of the initial test result must use a test that is different from the one used for the initial assessment. A reactive initial rapid test should be confirmed by either another type of rapid assay or an E/CIA that is based on a different antigen preparation and/or different test principle (e.g., indirect versus competitive), or a Western blot or a plasma HIV-1 RNA viral load.
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky performance status [KPS] >= 50)
* Life expectancy >= 12 weeks
* Hemoglobin >= 8 g/dL
* Absolute neutrophil count (ANC): >= 1,000 cells/mm^3 (1.0 x 10^9/L)
* Platelets: >= 75,000 cells/mm^3 (75.0 x 10^9/L)
* Total bilirubin: =< 1.5 times the upper limit of normal (ULN), unless the participant is receiving an antiretroviral drug known to be associated with increased bilirubin, in which case the direct fraction should be =< 2 times the ULN
* Serum aspartate aminotransferase (AST) serum glutamic-oxaloacetic transaminase (SGOT) / alanine aminotransferase (ALT) serum glutamate pyruvate transaminase (SGPT) =< 2.5 x ULN
* Estimated or measured creatinine clearance > 60 mL/minute (1.00 mL/s) (serum creatinine =< 2.0 mg/dL / 176.8 umol/L)
* Currently receiving local standard of care antiretroviral therapy (ART) for >= 12 weeks, with HIV viral load =< 400 copies/mL; participants are required to be on antiretroviral regimens that are in accordance with the current International AIDS Society guidelines concurrently with chemotherapy; the specific agents are at the discretion of the investigator and the use of investigational agents currently available on an expanded access basis is allowed
* A female of childbearing potential (FCBP) is a female who has achieved menarche at some point and who meets one of the following criteria: 1) has not undergone a hysterectomy or bilateral oophorectomy, or 2) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months), or 3) does not have a serum or plasma follicle stimulating hormone (FSH) > 40 mIU/mL and a history of amenorrhea x >= 1 year

  * FCBP must have a negative serum or urine pregnancy test with a sensitivity of at least 25 mIU/mL within 10-14 days prior to and again within 24 hours of starting pomalidomide and must either commit to continued abstinence from heterosexual intercourse or begin TWO acceptable methods of birth control, including one of the following highly effective, long-acting methods, DepoProvera, an intrauterine device (IUD), an implant*, or bilateral tubal ligation, if it can be verified that the procedure was performed, and one additional effective method AT THE SAME TIME, at least 28 days before she starts taking pomalidomide; FCBP must also agree to ongoing pregnancy testing
  * NOTE: Implants containing levonorgestrel and etonogestrel are prohibited in women receiving efavirenz, as drug interactions will render the implants ineffective
  * Men must agree to use a latex condom during sexual contact with a FCBP even if they have had a vasectomy
  * All participants must be counseled at a minimum of every 28 days about pregnancy precautions and risks of fetal exposure; serum or urine pregnancy testing will be repeated in FCBP, and must be negative, within 24 hours of starting each new cycle of pomalidomide
* Able to take aspirin (>= 81 mg) daily as prophylactic anticoagulation
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Participants who are receiving any other investigational agents
* Any prior use of thalidomide, lenalidomide, or pomalidomide
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to pomalidomide
* Visceral disease requiring cytotoxic chemotherapy (i.e., pulmonary KS, symptomatic gastrointestinal KS). KS-related lymphedema is permitted.
* Use of agents containing zidovudine (including Combivir and Trizivir) are prohibited; in order to be eligible, participants taking zidovudine must change to a different regimen at least 7 days prior to therapy initiation; changes to antiretroviral therapy (ART) therapy during the study may be made if medically necessary (toxicity, failure of regimen, etc.)

  * Use of medications or substances that are strong inhibitors of CYP1A2, which include amiodarone, cimetidine, fluoroquinolones (e.g., ciprofloxacin, enoxacin), fluvoxamine, and ticlopidine is prohibited
  * Use of erythropoietin is prohibited
  * Co-administration of corticosteroids greater than doses required for treatment of adrenal insufficiency is prohibited
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection for which the participant has not completed at least 14 days of therapy prior to study enrollment and/or is not clinically stable; symptomatic congestive heart failure; unstable angina pectoris; cardiac arrhythmia; or psychiatric illness/social situations that, in the opinion of the investigator, would limit compliance with study requirements
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with pomalidomide
* Specific KS therapy, including cytotoxic chemotherapy but not including ART, within the past 4 weeks
* Use of other anticancer treatments or agents within the past 4 weeks
* History of malignant tumors other than KS, unless:

  * In complete remission for >= 1 year, or
  * Completely resected basal cell carcinoma, or
  * In situ squamous cell carcinoma of the cervix or anus
* Grade >= 1 peripheral neuropathy
* History of myocardial infarction (MI), cerebrovascular accident, or venous or arterial thromboembolism, unless line-related thrombosis without embolus occurring within 1 year prior to study entry
* Known procoagulant disorder including prothrombin gene mutation 20210, antithrombin III deficiency, protein C deficiency, protein S deficiency and antiphospholipid syndrome but not including heterozygosity for the factor V Leiden mutation or the presence of a lupus anticoagulant in the absence of other criteria for the antiphospholipid syndrome
* Any condition, including the presence of current laboratory abnormalities or other factor that, in the opinion of the investigator, places the participant at unacceptable risk if they were to participate in the study or confounds the ability to interpret data from the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2021-04-26 (Actual); Primary Completion 2024-11-29 (Actual); Study Completion 2025-04-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan E. Krown, MD, Study Chair — AIDS Malignancy Consortium; Samantha Vogt, MD, MPH, Study Chair — Johns Hopkins University
Locations (3):
- Moi University School of Medicine, Eldoret, Kenya
- UNC Project Malawi, Lilongwe, Malawi
- Uganda Cancer Institute, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Pomalidomide)
Started | 26
Completed | 8
Not Completed | 18
Not completed — Adverse Event | 2
Not completed — Death | 1
Not completed — Withdrawal by Subject | 2
Not completed — Lack of Efficacy | 7
Not completed — Other | 6

BASELINE CHARACTERISTICS:
Population: Study participants who received study treatment
Arm/Group | Treatment (Pomalidomide)
Number analyzed (Participants) | 26
Age, Continuous [Median (Inter-Quartile Range); unit: years old] — Age at enrollment
  years old | 38.7 [31.2 to 42.7]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 24
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 26
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 26
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Malawi | 15
  Uganda | 5
  Kenya | 6
CD4 cells at baseline [Count of Participants; unit: Participants]
  CD4 cells >200/uL | 24
  CD4 cells <=200/uL | 2

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate
Description: The binomial proportion and its 95% exact confidence interval will be used to estimate the overall response rate.
Time Frame: Up to 48 weeks
Population: Study participants who received study treatment
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Treatment (Pomalidomide)
Number analyzed (Participants) | 26
proportion of participants | 0.577 [0.369 to 0.766]

2. Primary Outcome: Complete Response Rate
Description: The binomial proportion and its 95% exact confidence interval will be used to estimate the complete response rate
Time Frame: Up to 48 weeks
Population: Study participants who received study treatment
Measure: Number (95% Confidence Interval); unit: proportion of participants
Arm/Group | Treatment (Pomalidomide)
Number analyzed (Participants) | 26
proportion of participants | 0 [0 to 0.16]

3. Primary Outcome: Incidence of Adverse Events Defined as Grade 3 or Higher Toxicities Graded According to the National Cancer Institute Common Terminology Criteria for Adverse Events Version 5.0
Description: Incidence of Grade 3 or higher toxicity will be reported using percentage and corresponding 95% confidence interval. The binomial proportion and its 95% exact confidence interval will be used to estimate the proportion of participants who experience a grade 3 or higher toxicity.
Time Frame: Up to 1 year
Population: Study participants who received study treatment
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Pomalidomide)
Number analyzed (Participants) | 26
percentage of participants
  All adverse events | 57.7 [37.2 to 76]
  Treatment-related adverse events | 38.5 [20.9 to 59.3]

4. Secondary Outcome: Changes in CD4 T Cell Count
Description: Changes in CD4 counts and human immunodeficiency virus (HIV) viral load will be evaluated.
Time Frame: Baseline to up to 1 year
Population: Participants with CD4 measurement at baseline and 1 year
Measure: Mean (Standard Deviation); unit: CD4 T cell counts per mm^3
Arm/Group | Treatment (Pomalidomide)
Number analyzed (Participants) | 26
CD4 T cell counts per mm^3
  Baseline | 456 (247.5)
  Cycle 2 Day 1: number analyzed (Participants) | 23
  Cycle 2 Day 1 | 524.1 (194.2)
  Cycle4 Day 1: number analyzed (Participants) | 21
  Cycle4 Day 1 | 512.6 (251.5)
  Cycle 7 Day 1: number analyzed (Participants) | 8
  Cycle 7 Day 1 | 587.8 (327.3)
  Cycle 10 Day 1: number analyzed (Participants) | 8
  Cycle 10 Day 1 | 417.4 (203)
  Treatment Discontinuation: number analyzed (Participants) | 18
  Treatment Discontinuation | 484.6 (209)

5. Secondary Outcome: Changes in HIV Viral Load as Measured by HIV Quantitative Polymerase Chain Reaction
Description: Changes in CD4 counts and HIV viral load will be evaluated.
Time Frame: Baseline to up to 1 year
Population: Participants with HIV viral load measurement at baseline and 1 year
Measure: Mean (Standard Deviation); unit: HIV viral load copies per mL
Arm/Group | Treatment (Pomalidomide)
Number analyzed (Participants) | 26
HIV viral load copies per mL
  Baseline | 34.9 (62)
  Cycle 2 Day 1: number analyzed (Participants) | 25
  Cycle 2 Day 1 | 31.4 (33.5)
  Cycle 4 Day 1: number analyzed (Participants) | 22
  Cycle 4 Day 1 | 31.5 (24.8)
  Cycle 7 Day 1: number analyzed (Participants) | 10
  Cycle 7 Day 1 | 23.2 (27.8)
  Cycle 10 Day 1: number analyzed (Participants) | 8
  Cycle 10 Day 1 | 27.5 (21.2)
  Treatment Discontinuation: number analyzed (Participants) | 10
  Treatment Discontinuation | 39.1 (12.6)

6. Other Pre Specified Outcome: Changes in Serum Cytokine Levels as Measured by Luminex Assay
Description: General estimating equations will be used to evaluate changes in cytokine levels over time. Logistic regression analyses will be used to evaluate the association between cytokine levels and clinical response.
Time Frame: Baseline to up to 48 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Up to 1 year
Arm/Group | Treatment (Pomalidomide)
All-Cause Mortality (participants affected / at risk) | 3/26
Serious Adverse Events (participants affected / at risk) | 7/26
Other Adverse Events (participants affected / at risk) | 23/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pomalidomide) (N=26)
Blood and lymphatic system disorders (Blood and lymphatic system disorders) | 1 (1)
Eye disorders (Eye disorders) | 1 (1)
Eye pain (Eye disorders) | 1 (1)
Death NOS (General disorders) | 2 (2)
Fever (General disorders) | 1 (1)
Infections and infestations (Infections and infestations) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 1 (1)
Hyponatremia (Metabolism and nutrition disorders) | 1 (1)
Neoplasms benign, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Tumor hemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Social circumstances (Social circumstances) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment (Pomalidomide) (N=26)
Diarrhea (Gastrointestinal disorders) | 2 (2)
Conjunctivitis infective (Infections and infestations) | 2 (3)
Wound infection (Infections and infestations) | 2 (2)
Lymphocite count decreased (Investigations) | 2 (2)
Lymphocyte count increased (Investigations) | 3 (5)
Neutrophil count decreased (Investigations) | 14 (25)
Hyperkalemia (Metabolism and nutrition disorders) | 2 (2)
Hypoalbuminemia (Metabolism and nutrition disorders) | 2 (4)
Hypoglycemia (Metabolism and nutrition disorders) | 3 (4)
Myalgia (Musculoskeletal and connective tissue disorders) | 3 (3)
Peripheral sensory neuropathy (Nervous system disorders) | 4 (4)
Cough (Respiratory, thoracic and mediastinal disorders) | 6 (7)
Hypertension (Vascular disorders) | 11 (18)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-12-04): https://cdn.clinicaltrials.gov/large-docs/06/NCT03601806/Prot_SAP_000.pdf
  • Informed Consent Form (2023-12-04): https://cdn.clinicaltrials.gov/large-docs/06/NCT03601806/ICF_001.pdf